CLINICAL TRIAL: NCT07178886
Title: Breast Reconstruction and Radiotherapy: a Nationwide Cohort Study on Care Evaluation and Optimization
Brief Title: Breast Reconstruction and Radiotherapy
Acronym: CONRAD
Status: Recruiting | Type: Observational
Sponsor: Janine M. Simons MD PhD (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Maastro Clinic, The Netherlands (Other)
Responsible Party: Sponsor-Investigator, Janine M. Simons MD PhD, Principal Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: 10390032310055; 10390032310055 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-02-21; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Mastectomy; Radiotherapy; Reconstruction; Quality of life; Patient Reported Outcomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients, 18 years or older, treated with mastectomy and radiotherapy for breast cancer.: Adult patients with breast cancer (to be) treated with mastectomy who have an indication for radiotherapy and who may or may not undergo breast reconstruction will be included.
  The following treatments of interest will be identified:
  * "immediate breast reconstruction" (implant-based or autologous)
  * "delayed breast reconstruction" group (implant-based or autologous)
  * "no breast reconstruction" group

SUMMARY:
If the whole breast is removed because of breast cancer, several options for breast reconstruction are available. All these options have an increased complication risk if a patient has been or will be treated with radiotherapy. However, only a few high-quality studies addressed patient satisfaction and complication risks, both in terms of timing (prior to or after irradiation) and type of reconstruction (implant or own tissue). As radiotherapy indications expand and more patients desire a reconstruction, this is a progressively relevant issue. Through this nationwide prospective study, the investigators aim to identify the most ideal treatment strategy by comparing different reconstruction options in terms of patient reported outcomes (PROs), toxicity, oncological safety and costs. These results will enable improvement of shared decision-making and cost-effectiveness of breast reconstruction strategies in case of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with unilateral non-metastatic breast cancer
* (to be) Treated with mastectomy and to be treated with adjuvant radiotherapy
* Willing and able to provide written informed consent

Exclusion Criteria:

* History of DCIS or invasive breast cancer
* Previous thoracic radiotherapy treatment
* History of other malignancies (except for patients with basal or squamous cell skin cancer, in situ carcinoma of the cervix and patients who are disease-free at least 5 years following successful treatment for other malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with breast cancer (to be) treated with mastectomy who have an indication for radiotherapy and who may or may not undergo breast reconstruction will be included.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction at 1 year | From enrollment to one year follow-up after treatment.
  The primary objective is to assess patient reported outcomes at 1 year (after mastectomy), by means of the validated questionnaire BREAST-Q. With the BREAST-Q questionnaire, four domains will be evaluated (psychosocial well-being (score ranges from 10 to 50), physical well-being (score ranges from 10 to 30), sexual well-being (score ranges from 6 to 30) and satisfaction with breasts (score ranges from 4 to 16) and higher scores indicate better outcomes.
Patient quality of life at 1 year | From enrollment to one year follow-up after treatment.
  The primary objective is to assess patient reported outcomes at 1 year (after mastectomy), by means of the validated questionnaire EQ-5D-5L.
  The EQ-5D-5L questionnaire consists of two parts: the descriptive system, with a minimum value of 5 and maximum value of 25 (higher scores mean worse quality of life) and the visual analogue scale, with a minimum value of 0 and maximum value of 100 (higher scores mean better quality of life).

SECONDARY OUTCOMES:
Patient satisfaction at 3 and 5 years | From enrollment to 3 and 5 years follow-up after treatment.
  To assess patient reported outcomes at 3, and 5 years (after mastectomy), by means of the validated questionnaire BREAST-Q. With the BREAST-Q questionnaire, four domains will be evaluated (psychosocial well-being (score ranges from 10 to 50), physical well-being (score ranges from 10 to 30), sexual well-being (score ranges from 6 to 30) and satisfaction with breasts (score ranges from 4 to 16) and higher scores indicate better outcomes.
Patient quality of life at 3 and 5 years | From enrollment to 3 and 5 years follow-up after treatment.
  To assess patient reported outcomes at 3, and 5 years (after mastectomy), by means of the validated questionnaire EQ-5D-5L. The EQ-5D-5L questionnaire consists of two parts: the descriptive system, with a minimum value of 5 and maximum value of 25 (higher scores mean worse quality of life) and the visual analogue scale, with a minimum value of 0 and maximum value of 100 (higher scores mean better quality of life).
Complications prior to and following radiotherapy | From enrollment to end of study follow-up (i.e. 5 years after treatment).
  To assess complication rates prior to and after radiotherapy (e.g., total number of surgical reinterventions, reconstruction failure, capsular contracture, fibrosis, pain). Data on type of complications and complication rates (categorized as early (<90 days after surgery) or late (>90 days after surgery will be collected
Cost-effectiveness and consumption of medical care and materials. | Patients will be followed until 5 years after mastectomy (or 5 years after delayed breast reconstruction if applicable).
  The main outcomes of the economic evaluation will be the incremental cost-effectiveness per life-year gained and per quality-adjusted life-year gained. Primary care resource use (e.g., visits to the general practitioner, physiotherapist and home care) will be collected using the iMTA Medical Consumption Questionnaire (iMCQ), Productivity Cost Questionnaire (iPCQ) and Valuation of Informal Care Questionnaire (iVICQ) and administered at baseline (after surgery and before radiotherapy) and 3 months after surgery. Secondary care resource use (e.g., inpatient days, outpatient visits, RT and surgery procedures) will be obtained through DHD.
Time to adjuvant treatment (radiotherapy/systemic therapy). | Patients will be followed until 5 years after mastectomy (or 5 years after delayed breast reconstruction if applicable).
  To assess time to adjuvant oncologic treatment (radiotherapy/systemic therapy)
Breast cancer recurrence rates at 3, and 5 years | Patients will be followed until 5 years after mastectomy (or 5 years after delayed breast reconstruction if applicable).
  Regarding breast cancer recurrence and time-to-event analysis, any (invasive or in situ) local, regional or distant recurrence will be registered as a recurrence event. The locoregional recurrence rate is defined as the time from diagnosis to a local and/or regional recurrence. The distant recurrence rate is defined as the time from diagnosis to a distant recurrence.
Recurrence free interval, disease free survival and overall survival at 3 and 5 years. | Patients will be followed until 5 years after mastectomy (or 5 years after delayed breast reconstruction if applicable).
  The recurrence-free interval is defined as the time from diagnosis to any event related to breast cancer, including death from breast cancer. Disease free survival is defined as the time from diagnosis to any event related to breast cancer or death (irrespective of cause of death). Overall survival is defined as the time from diagnosis to death from any cause. Patients will be censored if lost to follow-up before 5 years of follow-up or if they are alive at 5 years follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Other scientist can contact the PI and request data. The purpose of the request should be provided in writing. If a data transfer is agreed upon, the data will be shared according to the Erasmus MC guidelines on data security and after a DTA has been signed by both parties.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared and reused only if and dependent on whether access to the data is approved by the Sponsor and PI of the study.
Access Criteria: The purpose of the request should be provided in writing. If a data transfer is agreed upon, the data will be shared according to the Erasmus MC guidelines on data security and after a DTA has been signed by both parties.